CLINICAL TRIAL: NCT03964831
Title: Visualization Study of the UWF (Ultra Wide-field) SLO (Scanning Laser Ophthalmoscope) RG (Red Green), AF (Autofluorescence), FA (Fluorescein Angiography) and ICG ( Indocyanine Green Fluorescence) Images Using the P200TxE (Indy) and P200DTx (California)
Brief Title: Study Comparing the P200TxE and P200DTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1035
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultra widefield image capture (Other)
  Interventions: Device: P200TxE; Device: P200DTx

INTERVENTIONS:
Device: P200TxE — The P200TxE ophthalmoscope provides widefield scanning laser ophthalmascope (SLO) fundus imaging.
Device: P200DTx — The P200DTx ophthalmoscope provides widefield scanning laser ophthalmascope (SLO) fundus imaging.

SUMMARY:
The study evaluates image quality between two devices.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site,
3. Subjects who agree to participate in the study;
4. Subjects diagnosed with retinal pathology. Example of pathologies may include but are not limited to Age-related Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Central Serous Retinopathy, and others as confirmed by the investigator;

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable images;

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Qualitative Image assessment | 6 months
  Results from a qualitative assessment of the clinical utility and image quality of the images from both devices will be assessed from a clinician questionnaire and three independent masked and qualified graders using a four point scale (0-3).
Safety Assessment from Adverse Events | 6 months
  Analysis of safety will be assessed through adverse events reported by the site and documented on each subject's case report form.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Ophthalmology Associates, San Antonio, Texas, United States